CLINICAL TRIAL: NCT00459225
Title: Iron Prophylaxis for Anemia in Infants With Cyanotic Congenital Heart Disease: An Open Label Trial
Brief Title: Iron Prophylaxis for Anemia in Infants With Cyanotic Congenital Heart Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty recruiting subjects
Sponsor: Emory University (Other)
Collaborators: Children's Healthcare of Atlanta (Other)
Responsible Party: Principal Investigator, William T. Mahle, MD, Director of Clinical Research, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00002287
Record Dates: First submitted 2007-04-10; First posted 2007-04-11 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Anemia
Keywords: Pediatrics; Cardiac Defect; Cardiac Surgery; Single Ventricle; Anemia; blood transfusions; red cell volume; red cell distribution; oral iron; ferrous sulfate; Congenital Cardiac Defects; Hemoglobin; Iron Deficiency
MeSH Terms: conditions — Anemia; Univentricular Heart; Heart Defects, Congenital; Iron Deficiencies | interventions — Iron-Dextran Complex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): The parent/guardian will be educated on the iron study and provided the opportunity to ask questions. If the parent/guardian chooses to participate in the study, the parent/guardian will give informed consent for the patient to be placed in either Group I or Group II, based upon guardian/parents' choice for participation in the iron arm of the study. Group I will be randomized in a 1:1 ratio in this open label trial to either receive or not receive iron. Group II will not receive iron but will be a participant in the study and follow the course of the non-iron randomized patients.
  Interventions: Drug: Iron (ferrous sulfate)
- 2 (No Intervention): Group II will not receive iron but will be a participant in the study and follow the course of the non-iron randomized patients.

INTERVENTIONS:
Drug: Iron (ferrous sulfate) — The subjects in the iron treatment arm of the study will receive 3 mg/kg of oral/enteral iron solution once a day beginning at the time of discharge until the pre-Glenn screening which is the endpoint of the study. The iron will be dispensed for the subjects upon discharge from the hospital. The subjects randomized to the no iron treatment arm and the patients in Group II of the study will not receive iron upon discharge. However, they may be started on iron therapy in an intent-to-treat anemia by their primary physician in which case this will serve as the endpoint of the study for these participants.
  Arms: 1

SUMMARY:
Anemia is a common disorder in infants with one working chamber of the heart that pumps blood. Anemia is when the level of healthy blood cells becomes too low. This may cause other health problems because red blood cells contain hemoglobin, which carries oxygen (needed for survival) to different parts of the body.

This study will look at the role of iron in preventing anemia in infants with one pumping chamber. The importance of iron therapy will be examined.

Hypothesis: Prophylactic use of iron in infants with single ventricle is effective in preventing anemia.

DETAILED DESCRIPTION:
At the beginning of the study, subjects will be randomized to two different groups. One group will receive iron every day for the next 4 months or so (up until their Glenn surgery); the other group will not receive any iron. Those in the iron treatment arm of the study will receive iron education at discharge from their first stage surgery (Norwood or BTS surgery) and will be given vials of iron to take home. A patient will receive a set amount of iron (dose will be 3 mg/kg) once a day. Weekly follow-up phone calls will be conducted by study personnel to re-calculate dose of iron for parents (based on weight) as well as check on the status of the research subject.

Group II will not receive iron but will be a participant in the study and follow the course of the non-iron randomized patients.

Blood samples will also be drawn at the same time as standard of care labs at two time points during the course of the study for both groups of patients. Blood for iron study labs will be drawn at 72 hours prior to discharge from the first stage surgery and at the pre-Glenn screening. A reticulocyte count test will also be done at the pre-Glenn screening. These lab tests look at the number of red blood cells in the body, the type of red blood cells, their ability to carry oxygen and the iron status of the research subject. Additionally, data will be collected on the CBC count, subject's age, weight, pulse oximetry, surgical history, transfusion history, iron levels and therapy, and hematological indices (Hgb, Hct, MCV, RDW, RBC count, and reticulocyte count), as well as peripheral blood smear. Feeding history will be carefully documented. Descriptive demographic data and underlying diagnosis will be collected, along with all the above variables defined.

The hemoglobin and iron levels at the time of pre-Glenn labs will be compared to those at the start of the study. The importance of iron therapy will be examined.

Iron is a readily available medicine for both the prevention and treatment of anemia. If this simple cost-effective medicine can decrease the prevalence of anemia in these infants, it may result in more oxygen to the body's tissues and areas, less stress on the single pumping chamber of the heart and it may also improve their overall growth and development.

1. Primary Aim - To achieve a higher hemoglobin level at time of second stage surgery (Glenn procedure).
2. Secondary Aims - To obtain the following outcomes:

   1. Increased ferritin levels
   2. Decreased interval blood transfusions
   3. Normal MCV (red cell volume) and RDW (red cell distribution)

ELIGIBILITY:
Inclusion Criteria:

* Single ventricle physiology (hypoplastic left heart syndrome [HLHS], tricuspid atresia, double inlet left ventricle [DILV], some double outlet right ventricle [DORV], heterotaxy, etc.)
* Age less than or equal to 2 months
* Saturations less than or equal to 90%
* Tolerating enteral feeds
* Informed consent being obtained

Exclusion Criteria:

* Age > 2 months
* Saturations > 90%
* Total parenteral nutrition
* Chronic kidney disease
* Prior iron therapy
* Hemolytic anemia

Max Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2007-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Complete blood count, Iron study labs (ferritin, Total Iron Binding Capacity, and Iron lab) 72 hours prior to discharge following neonatal surgery | Discharge from hospital
Hemoglobin and Hematocrit at pre-Glenn catheterization | Will be assessed at the pre-Genn catheterization
Complete Blood count, Iron study labs, and Reticulocyte count at pre-glenn screening | Will be assessed at the pre-glenn screening

SECONDARY OUTCOMES:
feeding regimen and transfusion history at 72 hours prior to discharge from neonatal surgery, at pre-Glenn catheterization, and at pre-Glenn screening | Will be assessed at the time of discharge, pre-Glenn catheterization and screening.

CONTACTS AND LOCATIONS:
Overall Officials: William Mahle, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States

REFERENCES:
- [Background] Kaemmerer H, Fratz S, Braun SL, Koelling K, Eicken A, Brodherr-Heberlein S, Pietrzik K, Hess J. Erythrocyte indexes, iron metabolism, and hyperhomocysteinemia in adults with cyanotic congenital cardiac disease. Am J Cardiol. 2004 Sep 15;94(6):825-8. doi: 10.1016/j.amjcard.2004.06.014. PMID 15374802
- [Background] Perloff JK, Rosove MH, Child JS, Wright GB. Adults with cyanotic congenital heart disease: hematologic management. Ann Intern Med. 1988 Sep 1;109(5):406-13. doi: 10.7326/0003-4819-109-5-406. PMID 3044212
- [Background] Perloff JK. Systemic complications of cyanosis in adults with congenital heart disease. Hematologic derangements, renal function, and urate metabolism. Cardiol Clin. 1993 Nov;11(4):689-99. PMID 8252568
- [Background] Felker GM, Shaw LK, Stough WG, O'Connor CM. Anemia in patients with heart failure and preserved systolic function. Am Heart J. 2006 Feb;151(2):457-62. doi: 10.1016/j.ahj.2005.03.056. PMID 16442914
- [Background] Dallman PR, Siimes MA, Stekel A. Iron deficiency in infancy and childhood. Am J Clin Nutr. 1980 Jan;33(1):86-118. doi: 10.1093/ajcn/33.1.86. No abstract available. PMID 6986756